CLINICAL TRIAL: NCT02458638
Title: An Open-Label, Multicohort, Phase II Study of Atezolizumab in Advanced Solid Tumors
Brief Title: A Study of Atezolizumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO29518; 2015-000269-30 (EudraCT Number)
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atezolizumab (Experimental): The dose of atezolizumab in this study will be 1200 milligrams (mg) administered by intravenous (IV) infusion on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody — Atezolizumab will be given as IV infusion over 60 minutes on Day 1 of Cycle 1, then over 30 minutes (as tolerated) on Day 1 of each subsequent 3-week cycle.
  Other Names: Tecentriq

SUMMARY:
The primary efficacy objective for this study is to evaluate non-progression rate (NPR) at 18 weeks in participants with advanced solid tumors treated with atezolizumab, defined as the percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1, or according to disease-specific criteria for prostate cancer and malignant pleural mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented advanced solid tumors that meet protocol-defined cohort specifications, have progressive disease at study entry, and have received at least one line of prior systemic therapy or for which no alternative therapy to prolong survival exists
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (preferred) or in freshly cut and unstained slides (exceptional cases) with an associated pathology report for central testing
* Measurable disease as defined by RECIST v1.1 or disease-specific criteria for prostate cancer and malignant pleural mesothelioma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Negative serum pregnancy test result within 14 days prior to study drug among women of childbearing potential
* Life expectancy > 3 months

Exclusion Criteria:

* Malignancies other than disease under study within 5 years prior to Day 1 of Cycle 1 except those with a negligible risk of metastasis or death
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures >/=1 time per month
* History of asymptomatic or symptomatic central nervous system (CNS) metastasis
* Leptomeningeal disease
* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated but without evidence that disease has been clinically stable for >/=2 weeks prior to Day 1 of Cycle 1
* Pregnant and lactating women
* Significant cardiovascular disease within 3 months prior to Day 1 of Cycle 1
* Severe infection within 4 weeks prior to Day 1 of Cycle 1
* Oral or IV antibiotics within 2 weeks prior to Day 1 of Cycle 1
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation
* History of autoimmune disease except treated/stable hypothyroidism, Type 1 diabetes mellitus, and protocol-specified dermatologic conditions
* Active tuberculosis
* Signs or symptoms of infection within 2 weeks prior to Day 1 of Cycle 1
* Prior treatment with cluster of differentiation (CD) 137 agonists or immune checkpoint blockade therapies, or anti-programmed cell death-1 (PD-1) or anti-PD-L1 therapeutic antibodies
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to Day 1 of Cycle 1, or anticipated requirement for systemic immunosuppressive medications during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- United States (5):
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Sarah Cannon Cancer Center and Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Austria (2):
  - LKH-UNIV. KLINIKUM GRAZ; Klinische Abteilung für Onkologie, Graz
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Chemotherapie & Infektionskrankhei, Vienna
- Brazil (3):
  - INCA 1- Instituto Nacional de Câncer X, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
- Denmark (3):
  - Aarhus Universitetshospital; Kræftafdelingen, Aarhus N
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Odense Universitetshospital, Onkologisk Afdeling, Klinisk Forsknings Enhed, Odense C
- Helsinki University Central Hospital; Dept of Oncology, Helsinki, Finland
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Hopital Saint Louis, Service D Oncologie Medicale, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Uniklinik-Eppendorf; Zentren F. Innere Medizin-Klinik U. Poliklinik, Hamburg
  - Universitatsklinik Heidelberg; Universitätshautklinik und Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
- Ireland (2):
  - St Vincent'S Uni Hospital; Medical Oncology, Dublin
  - St James' Hospital; Cancer Clinical Trials Office, Dublin
- Italy (3):
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
- Netherlands (3):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Norway (2):
  - Haukeland Universitetssjukehus; Klinisk forskningspost, Bergen
  - Oslo Universitetssykehus HF; Radiumhospitalet, Oslo
- Poland (3):
  - Centrum Onkologii w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne; Klinika Onkologii i Radioterapii, Gdansk
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie; Klinika Now. Tkanek Miekkich,Kosci i Czer., Warsaw
- Russia (2):
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg
- Spain (2):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
- Switzerland (2):
  - Freiburger Spital; Onkologie, Fribourg
  - Kantonsspital St. Gallen; Onkologie/Hämatologie, Sankt Gallen
- Turkey (Türkiye) (4):
  - Trakya University Medical Faculty, Edirne
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - Prof. Dr. Cemil Tascioglu City Hospital; Med Onc, Istanbul
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara
- United Kingdom (2):
  - Clatterbridge Cancer Centre, Bebington
  - Southampton General Hospital; Medical Oncology, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tabernero J, Andre F, Blay JY, Bustillos A, Fear S, Ganta S, Jaeger D, Maio M, Mileshkin L, Melero I. Phase II multicohort study of atezolizumab monotherapy in multiple advanced solid cancers. ESMO Open. 2022 Apr;7(2):100419. doi: 10.1016/j.esmoop.2022.100419. Epub 2022 Mar 16. PMID 35305400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 47 sites in 18 countries: Austria, Brazil, Canada, Denmark, Finland, France, Germany, Ireland, Italy, Netherlands, Norway, Poland, Russian Federation, Spain, Switzerland, Turkey, United Kingdom and United States.
Pre-assignment Details: Participants with advanced solid tumors were eligible to enroll in the study.
Groups:
- Atezolizumab: Atezolizumab 1200 milligrams (mg) was administered by intravenous (IV) infusion on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Atezolizumab
Started | 474
Completed | 15
Not Completed | 459
Not completed — Death | 309
Not completed — End of Cohort/End of Study | 67
Not completed — Lost to Follow-up | 31
Not completed — Other Reasons | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 47

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab
Number analyzed (Participants) | 474
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233
  Male | 241
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18
  Asian | 1
  Black or African American | 5
  Native Hawaiian Other Pacific Island | 4
  White | 406
  Unknown race | 37
  Not Reported In France | 2
  Not Available | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 383
  Not reported | 34
  Unknown | 17

OUTCOME MEASURES:

1. Primary Outcome: Non-progression Rate (NPR) at 18 Weeks
Description: NPR was defined as the percentage of participants with complete response (CR), partial response (PR) or stable disease (SD) as assessed by the Investigator according to Response Evaluation Criteria in Solid Tumors (RECIST), v1.1 or for malignant pleural mesothelioma according to Malignant Pleural Mesothelioma Response Evaluation Criteria. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions in the absence of CR. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD: At least a 20% increase in the sum of diameters of all target and all new measurable lesions. For prostate cancer according to Prostate Response Evaluation Criteria. CR: PSA <5 ng/ml measured twice at least 3 weeks apart or PSA response: PSA < 50% of the PSA reference value occurring at any time after treatment was initiated.
Time Frame: At Week 18
Population: Efficacy analysis set included all eligible and evaluable participants. A participant was considered evaluable if they received study drug, had a baseline tumor assessment and at least one tumor assessment post-baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population | 26.8 [22.7 to 31.2]
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 44.4 [25.5 to 64.7]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 29.6 [13.8 to 50.2]
  High Microsatellite Instability (MSI-H) or Mismatch Repair (MMR) Deficient Colorectal Cancer: number analyzed (Participants) | 10
  High Microsatellite Instability (MSI-H) or Mismatch Repair (MMR) Deficient Colorectal Cancer | 40.0 [12.2 to 73.8]
  Breast Cancer Type 1/2 Susceptibility Protein (BRCA) Mutated Ovarian Cancer: number analyzed (Participants) | 15
  Breast Cancer Type 1/2 Susceptibility Protein (BRCA) Mutated Ovarian Cancer | 26.7 [7.8 to 55.1]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 0 [0 to 26.5]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 7.7 [0.2 to 36.0]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 17.6 [3.8 to 43.4]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 20.0 [4.3 to 48.1]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 0 [0 to 28.5]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 23.1 [9.0 to 43.6]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 25.0 [3.2 to 65.1]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 45.5 [16.7 to 76.6]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 16.7 [2.1 to 48.4]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 38.5 [13.9 to 68.4]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 42.9 [17.7 to 71.1]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 15.4 [1.9 to 45.4]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 6.7 [0.2 to 31.9]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 54.5 [23.4 to 83.3]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 28.6 [3.7 to 71.0]
  Gastric/Gastro-esophageal (GE) Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/Gastro-esophageal (GE) Junction Adenocarcinoma | 21.4 [4.7 to 50.8]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 7.1 [0.2 to 33.9]
  Estrogen Receptor (ER)+/Human EGF Receptor 2 (HER2)- Hypermutated Metastatic Breast Cancer (MBC): number analyzed (Participants) | 12
  Estrogen Receptor (ER)+/Human EGF Receptor 2 (HER2)- Hypermutated Metastatic Breast Cancer (MBC) | 8.3 [0.2 to 38.5]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 76.9 [46.2 to 95.0]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 41.7 [15.2 to 72.3]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 58.3 [27.7 to 84.8]
  Poorly Differentiated Grade (excluding small cell lung cancer [SCLC]): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding small cell lung cancer [SCLC]) | 25.0 [5.5 to 57.2]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 33.3 [4.3 to 77.7]
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 0 [0 to 60.2]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 18.2 [2.3 to 51.8]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 40.0 [12.2 to 73.8]

2. Secondary Outcome: NPR at 24 Weeks
Description: as for outcome 1
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population | 22.4 [18.6 to 26.6]
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 40.7 [22.4 to 61.2]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 22.2 [8.6 to 42.3]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 40.0 [12.2 to 73.8]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 20.0 [4.3 to 48.1]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 0 [0 to 26.5]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 7.7 [0.2 to 36.0]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 11.8 [1.5 to 36.4]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 13.3 [1.7 to 40.5]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 0 [0 to 28.5]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 23.1 [9.0 to 43.6]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 25.0 [3.2 to 65.1]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 45.5 [16.7 to 76.6]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 0 [0 to 26.5]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 23.1 [5.0 to 53.8]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 28.6 [8.4 to 58.1]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 7.7 [0.2 to 36.0]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 6.7 [0.2 to 31.9]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 54.5 [23.4 to 83.3]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 28.6 [3.7 to 71.0]
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 7.1 [0.2 to 33.9]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 7.1 [0.2 to 33.9]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 8.3 [0.2 to 38.5]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 76.9 [46.2 to 95.0]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 33.3 [9.9 to 65.1]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 58.3 [27.7 to 84.8]
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 16.7 [2.1 to 48.4]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 16.7 [0.4 to 64.1]
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 0 [0 to 60.2]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 18.2 [2.3 to 51.8]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 30.0 [6.7 to 65.2]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with CR or PR as assessed by the investigator using RECIST v1.1 or Malignant Pleural Mesothelioma Response Evaluation Criteria. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions, taking as reference the baseline sum of diameters, in the absence of CR. For prostate cancer according to Prostate Response Evaluation Criteria. CR: PSA <5 ng/ml measured twice at least 3 weeks apart or PSA response: PSA < 50% of the PSA reference value occurring at any time after treatment was initiated.
Time Frame: Baseline up to 4.5 years (assessed every 6 weeks for first 24 weeks and thereafter every 12 weeks up to loss of clinical benefit, withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population | 7.4 [5.1 to 10.3]
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 14.8 [4.2 to 33.7]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 7.4 [0.9 to 24.3]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 0 [0 to 30.8]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 13.3 [1.7 to 40.5]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 0 [0 to 26.5]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 0 [0 to 24.7]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 5.9 [0.1 to 28.7]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 0 [0 to 21.8]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 0 [0 to 28.5]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 7.7 [0.9 to 25.1]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 12.5 [0.3 to 52.7]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 9.1 [0.2 to 41.3]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 0 [0 to 26.5]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 7.7 [0.2 to 36.0]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 14.3 [1.8 to 42.8]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 0 [0 to 24.7]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 0 [0 to 21.8]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 9.1 [0.2 to 41.3]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 0 [0 to 41.0]
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 7.1 [0.2 to 33.9]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 0 [0 to 23.2]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 8.3 [0.2 to 38.5]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 38.5 [13.9 to 68.4]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 8.3 [0.2 to 38.5]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 0 [0 to 26.5]
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 16.7 [2.1 to 48.4]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 16.7 [0.4 to 64.1]
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 0 [0 to 60.2]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 9.1 [0.2 to 41.3]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 20.0 [2.5 to 55.6]

4. Secondary Outcome: Percentage of Participants by Best Overall Response (BOR)
Description: BOR was based on RECIST v1.1, Malignant Pleural Mesothelioma Response Evaluation Criteria or Prostate Response Evaluation Criteria. For an individual participant BOR was obtained as follows: 1) CR: overall tumor response assessment of CR at 2 consecutive visits at least 28 days apart. 2) PR: overall tumor response assessment of PR or CR at 2 consecutive visits at least 28 days apart without being a CR. 3) SD: overall tumor response assessment of SD, PR, or CR at one or more visits at least 42 days after start of study treatment, but was not a confirmed CR or PR. 4) PD: an overall tumor response assessment of PD at any visit, and did not meet the criteria for a BOR of CR, PR or SD. 5) Missing: an assessment of SD, PR or CR in the first 42 days after start of study treatment and no further tumor assessments thereafter.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population: CR | 0.7
  Overall Population: PR | 6.7
  Overall Population: SD | 36.3
  Overall Population: PD | 53.3
  Overall Population: Missing | 3.0
  Cervical Cancer: CR: number analyzed (Participants) | 27
  Cervical Cancer: CR | 3.7
  Cervical Cancer: PR: number analyzed (Participants) | 27
  Cervical Cancer: PR | 11.1
  Cervical Cancer: SD: number analyzed (Participants) | 27
  Cervical Cancer: SD | 40.7
  Cervical Cancer: PD: number analyzed (Participants) | 27
  Cervical Cancer: PD | 40.7
  Cervical Cancer: Missing: number analyzed (Participants) | 27
  Cervical Cancer: Missing | 3.7
  Nasopharyngeal Carcinoma: CR: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: CR | 0
  Nasopharyngeal Carcinoma: PR: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: PR | 7.4
  Nasopharyngeal Carcinoma: SD: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: SD | 44.4
  Nasopharyngeal Carcinoma: PD: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: PD | 48.1
  Nasopharyngeal Carcinoma: Missing: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: Missing | 0
  MSI-H or MMR Deficient Colorectal Cancer: CR: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: CR | 0
  MSI-H or MMR Deficient Colorectal Cancer: PR: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: PR | 0
  MSI-H or MMR Deficient Colorectal Cancer: SD: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: SD | 40.0
  MSI-H or MMR Deficient Colorectal Cancer: PD: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: PD | 50.0
  MSI-H or MMR Deficient Colorectal Cancer: Missing: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: Missing | 10.0
  BRCA Mutated Ovarian Cancer: CR: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: CR | 0
  BRCA Mutated Ovarian Cancer: PR: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: PR | 13.3
  BRCA Mutated Ovarian Cancer: SD: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: SD | 33.3
  BRCA Mutated Ovarian Cancer: PD: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: PD | 46.7
  BRCA Mutated Ovarian Cancer: Missing: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: Missing | 6.7
  BRCA Mutated Breast Cancer: CR: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: CR | 0
  BRCA Mutated Breast Cancer: PR: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: PR | 0
  BRCA Mutated Breast Cancer: SD: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: SD | 8.3
  BRCA Mutated Breast Cancer: PD: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: PD | 91.7
  BRCA Mutated Breast Cancer: Missing: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: Missing | 0
  Liposarcoma: CR: number analyzed (Participants) | 13
  Liposarcoma: CR | 0
  Liposarcoma: PR: number analyzed (Participants) | 13
  Liposarcoma: PR | 0
  Liposarcoma: SD: number analyzed (Participants) | 13
  Liposarcoma: SD | 30.8
  Liposarcoma: PD: number analyzed (Participants) | 13
  Liposarcoma: PD | 61.5
  Liposarcoma: Missing: number analyzed (Participants) | 13
  Liposarcoma: Missing | 7.7
  Leiomyosarcoma: CR: number analyzed (Participants) | 17
  Leiomyosarcoma: CR | 0
  Leiomyosarcoma: PR: number analyzed (Participants) | 17
  Leiomyosarcoma: PR | 5.9
  Leiomyosarcoma: SD: number analyzed (Participants) | 17
  Leiomyosarcoma: SD | 17.6
  Leiomyosarcoma: PD: number analyzed (Participants) | 17
  Leiomyosarcoma: PD | 64.7
  Leiomyosarcoma: Missing: number analyzed (Participants) | 17
  Leiomyosarcoma: Missing | 11.8
  Gastrointestinal Stromal Tumor (GIST): CR: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): CR | 0
  Gastrointestinal Stromal Tumor (GIST): PR: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): PR | 0
  Gastrointestinal Stromal Tumor (GIST): SD: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): SD | 33.3
  Gastrointestinal Stromal Tumor (GIST): PD: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): PD | 66.7
  Gastrointestinal Stromal Tumor (GIST): Missing: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): Missing | 0
  Undifferentiated Pleomorphic Sarcoma: CR: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: CR | 0
  Undifferentiated Pleomorphic Sarcoma: PR: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: PR | 0
  Undifferentiated Pleomorphic Sarcoma: SD: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: SD | 9.1
  Undifferentiated Pleomorphic Sarcoma: PD: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: PD | 90.9
  Undifferentiated Pleomorphic Sarcoma: Missing: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: Missing | 0
  Known Translocation-Related Sarcomas: CR: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: CR | 0
  Known Translocation-Related Sarcomas: PR: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: PR | 7.7
  Known Translocation-Related Sarcomas: SD: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: SD | 34.6
  Known Translocation-Related Sarcomas: PD: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: PD | 53.8
  Known Translocation-Related Sarcomas: Missing: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: Missing | 3.8
  Radiation Induced Sarcoma: CR: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: CR | 0
  Radiation Induced Sarcoma: PR: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: PR | 12.5
  Radiation Induced Sarcoma: SD: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: SD | 12.5
  Radiation Induced Sarcoma: PD: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: PD | 75.0
  Radiation Induced Sarcoma: Missing: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: Missing | 0
  Osteosarcoma: CR: number analyzed (Participants) | 11
  Osteosarcoma: CR | 0
  Osteosarcoma: PR: number analyzed (Participants) | 11
  Osteosarcoma: PR | 9.1
  Osteosarcoma: SD: number analyzed (Participants) | 11
  Osteosarcoma: SD | 36.4
  Osteosarcoma: PD: number analyzed (Participants) | 11
  Osteosarcoma: PD | 54.5
  Osteosarcoma: Missing: number analyzed (Participants) | 11
  Osteosarcoma: Missing | 0
  Chondrosarcoma: CR: number analyzed (Participants) | 12
  Chondrosarcoma: CR | 0
  Chondrosarcoma: PR: number analyzed (Participants) | 12
  Chondrosarcoma: PR | 0
  Chondrosarcoma: SD: number analyzed (Participants) | 12
  Chondrosarcoma: SD | 41.7
  Chondrosarcoma: PD: number analyzed (Participants) | 12
  Chondrosarcoma: PD | 58.3
  Chondrosarcoma: Missing: number analyzed (Participants) | 12
  Chondrosarcoma: Missing | 0
  Pleural Mesothelioma: CR: number analyzed (Participants) | 13
  Pleural Mesothelioma: CR | 0
  Pleural Mesothelioma: PR: number analyzed (Participants) | 13
  Pleural Mesothelioma: PR | 7.7
  Pleural Mesothelioma: SD: number analyzed (Participants) | 13
  Pleural Mesothelioma: SD | 61.5
  Pleural Mesothelioma: PD: number analyzed (Participants) | 13
  Pleural Mesothelioma: PD | 30.8
  Pleural Mesothelioma: Missing: number analyzed (Participants) | 13
  Pleural Mesothelioma: Missing | 0
  Peritoneal Mesothelioma: CR: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: CR | 0
  Peritoneal Mesothelioma: PR: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: PR | 14.3
  Peritoneal Mesothelioma: SD: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: SD | 42.9
  Peritoneal Mesothelioma: PD: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: PD | 42.9
  Peritoneal Mesothelioma: Missing: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: Missing | 0
  Cholangiocarcinoma/Cancer of the Biliary Tract: CR: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: CR | 0
  Cholangiocarcinoma/Cancer of the Biliary Tract: PR: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: PR | 0
  Cholangiocarcinoma/Cancer of the Biliary Tract: SD: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: SD | 53.8
  Cholangiocarcinoma/Cancer of the Biliary Tract: PD: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: PD | 46.2
  Cholangiocarcinoma/Cancer of the Biliary Tract: Missing: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: Missing | 0
  Anaplastic Thyroid Cancer (TC): CR: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): CR | 0
  Anaplastic Thyroid Cancer (TC): PR: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): PR | 0
  Anaplastic Thyroid Cancer (TC): SD: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): SD | 13.3
  Anaplastic Thyroid Cancer (TC): PD: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): PD | 73.3
  Anaplastic Thyroid Cancer (TC): Missing: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): Missing | 13.3
  Follicular or Papillary Thyroid Cancer (TC): CR: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): CR | 0
  Follicular or Papillary Thyroid Cancer (TC): PR: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): PR | 9.1
  Follicular or Papillary Thyroid Cancer (TC): SD: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): SD | 72.7
  Follicular or Papillary Thyroid Cancer (TC): PD: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): PD | 18.2
  Follicular or Papillary Thyroid Cancer (TC): Missing: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): Missing | 0
  Medullary/Follicular/Papillary TC: CR: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: CR | 0
  Medullary/Follicular/Papillary TC: PR: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: PR | 0
  Medullary/Follicular/Papillary TC: SD: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: SD | 42.9
  Medullary/Follicular/Papillary TC: PD: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: PD | 42.9
  Medullary/Follicular/Papillary TC: Missing: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: Missing | 14.3
  Gastric/GE Junction Adenocarcinoma: CR: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: CR | 0
  Gastric/GE Junction Adenocarcinoma: PR: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: PR | 7.1
  Gastric/GE Junction Adenocarcinoma: SD: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: SD | 21.4
  Gastric/GE Junction Adenocarcinoma: PD: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: PD | 57.1
  Gastric/GE Junction Adenocarcinoma: Missing: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: Missing | 14.3
  Malignant Germ Cell Tumors: CR: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: CR | 0
  Malignant Germ Cell Tumors: PR: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: PR | 0
  Malignant Germ Cell Tumors: SD: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: SD | 35.7
  Malignant Germ Cell Tumors: PD: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: PD | 64.3
  Malignant Germ Cell Tumors: Missing: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: Missing | 0
  ER+/HER2- Hypermutated MBC: CR: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: CR | 0
  ER+/HER2- Hypermutated MBC: PR: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: PR | 8.3
  ER+/HER2- Hypermutated MBC: SD: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: SD | 8.3
  ER+/HER2- Hypermutated MBC: PD: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: PD | 83.3
  ER+/HER2- Hypermutated MBC: Missing: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: Missing | 0
  Thymoma: CR: number analyzed (Participants) | 13
  Thymoma: CR | 0
  Thymoma: PR: number analyzed (Participants) | 13
  Thymoma: PR | 38.5
  Thymoma: SD: number analyzed (Participants) | 13
  Thymoma: SD | 46.2
  Thymoma: PD: number analyzed (Participants) | 13
  Thymoma: PD | 7.7
  Thymoma: Missing: number analyzed (Participants) | 13
  Thymoma: Missing | 7.7
  Thymic cancer: CR: number analyzed (Participants) | 12
  Thymic cancer: CR | 0
  Thymic cancer: PR: number analyzed (Participants) | 12
  Thymic cancer: PR | 8.3
  Thymic cancer: SD: number analyzed (Participants) | 12
  Thymic cancer: SD | 50.0
  Thymic cancer: PD: number analyzed (Participants) | 12
  Thymic cancer: PD | 41.7
  Thymic cancer: Missing: number analyzed (Participants) | 12
  Thymic cancer: Missing | 0
  Low/Intermediate Grade Carcinoid: CR: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: CR | 0
  Low/Intermediate Grade Carcinoid: PR: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: PR | 0
  Low/Intermediate Grade Carcinoid: SD: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: SD | 100.0
  Low/Intermediate Grade Carcinoid: PD: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: PD | 0
  Low/Intermediate Grade Carcinoid: Missing: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: Missing | 0
  Poorly Differentiated Grade (excluding SCLC): CR: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): CR | 0
  Poorly Differentiated Grade (excluding SCLC): PR: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): PR | 16.7
  Poorly Differentiated Grade (excluding SCLC): SD: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): SD | 16.7
  Poorly Differentiated Grade (excluding SCLC): PD: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): PD | 66.7
  Poorly Differentiated Grade (excluding SCLC): Missing: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): Missing | 0
  Head and Neck Squamous Cell Carcinoma: CR: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: CR | 16.7
  Head and Neck Squamous Cell Carcinoma: PR: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: PR | 0
  Head and Neck Squamous Cell Carcinoma: SD: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: SD | 33.3
  Head and Neck Squamous Cell Carcinoma: PD: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: PD | 50.0
  Head and Neck Squamous Cell Carcinoma: Missing: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: Missing | 0
  Penile Cancer: CR: number analyzed (Participants) | 4
  Penile Cancer: CR | 0
  Penile Cancer: PR: number analyzed (Participants) | 4
  Penile Cancer: PR | 0
  Penile Cancer: SD: number analyzed (Participants) | 4
  Penile Cancer: SD | 50.0
  Penile Cancer: PD: number analyzed (Participants) | 4
  Penile Cancer: PD | 50.0
  Penile Cancer: Missing: number analyzed (Participants) | 4
  Penile Cancer: Missing | 0
  Anal Cancer: CR: number analyzed (Participants) | 11
  Anal Cancer: CR | 9.1
  Anal Cancer: PR: number analyzed (Participants) | 11
  Anal Cancer: PR | 0
  Anal Cancer: SD: number analyzed (Participants) | 11
  Anal Cancer: SD | 36.4
  Anal Cancer: PD: number analyzed (Participants) | 11
  Anal Cancer: PD | 54.5
  Anal Cancer: Missing: number analyzed (Participants) | 11
  Anal Cancer: Missing | 0
  Known MSI High or MMR Deficient Tumors: CR: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: CR | 0
  Known MSI High or MMR Deficient Tumors: PR: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: PR | 20.0
  Known MSI High or MMR Deficient Tumors: SD: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: SD | 40.0
  Known MSI High or MMR Deficient Tumors: PD: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: PD | 40.0
  Known MSI High or MMR Deficient Tumors: Missing: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: Missing | 0

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with CR, PR, or SD according to RECIST v1.1, Malignant Pleural Mesothelioma Response Evaluation Criteria or Prostate Response Evaluation Criteria lasting for >/=6 weeks. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions in the absence of CR. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD: At least a 20% increase in the sum of diameters of all target and all new measurable lesions. For prostate cancer: CR: PSA <5 ng/ml measured twice at least 3 weeks apart or PSA response: PSA < 50% of the PSA reference value occurring at any time after treatment was initiated.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population | 43.6 [38.9 to 48.5]
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 55.6 [35.3 to 74.5]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 51.9 [31.9 to 71.3]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 40.0 [12.2 to 73.8]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 46.7 [21.3 to 73.4]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 8.3 [0.2 to 38.5]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 30.8 [9.1 to 61.4]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 23.5 [6.8 to 49.9]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 33.3 [11.8 to 61.6]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 9.1 [0.2 to 41.3]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 42.3 [23.4 to 63.1]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 25.0 [3.2 to 65.1]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 45.5 [16.7 to 76.6]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 41.7 [15.2 to 72.3]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 69.2 [38.6 to 90.9]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 57.1 [28.9 to 82.3]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 53.8 [25.1 to 80.8]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 13.3 [1.7 to 40.5]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 81.8 [48.2 to 97.7]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 42.9 [9.9 to 81.6]
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 28.6 [8.4 to 58.1]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 35.7 [12.8 to 64.9]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 16.7 [2.1 to 48.4]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 84.6 [54.6 to 98.1]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 58.3 [27.7 to 84.8]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 100.0 [73.5 to 100.0]
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 33.3 [9.9 to 65.1]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 50.0 [11.8 to 88.2]
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 50.0 [6.8 to 93.2]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 45.5 [16.7 to 76.6]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 60.0 [26.2 to 87.8]

6. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR, based on RECIST v1.1, was defined as the time from the first occurrence of a documented objective response (CR or PR) to the time of progression or death from any cause, whichever occurred first. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions in the absence of CR. PD: At least a 20% increase in the sum of diameters of all target and all new measurable lesions. As pre-specified in the Statistical Analysis Plan (SAP) DOR was not analyzed if there were less than 4 participants available for the analysis.
Time Frame: as for outcome 3
Population: Efficacy analysis set included all eligible and evaluable participants. A participant was considered evaluable if they received study drug, had a baseline tumor assessment and at least one tumor assessment post-baseline. As pre-specified in the SAP DOR was not analyzed if there were less than 4 participants available for the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 14
months
  Cervical Cancer: number analyzed (Participants) | 4
  Cervical Cancer | 12.6 [3.0 to 15.2]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 4
  Nasopharyngeal Carcinoma | NA [1.1 to NA] — Median and upper limit of CI were not reached due to low number of participants with events.
  Thymoma: number analyzed (Participants) | 6
  Thymoma | 19.0 [1.5 to NA] — Upper limit of CI was not reached due to low number of participants with events.

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS, based on RECIST v1.1, was defined as the time from the first day of study treatment to the first occurrence of disease progression or death from any cause, whichever occurred first. PD: At least a 20% increase in the sum of diameters of all target and all new measurable lesions.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 397
months
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 4.14 [1.31 to 8.34]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 3.15 [1.35 to 4.60]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 1.51 [0.72 to 10.97]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 2.73 [1.45 to 4.01]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 1.38 [0.99 to 1.54]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 1.51 [1.25 to 4.70]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 2.69 [1.28 to 3.12]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 1.41 [1.15 to 2.79]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 1.31 [1.25 to 1.35]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 2.73 [1.38 to 5.42]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 1.43 [1.25 to 14.39]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 2.96 [1.28 to 16.69]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 1.87 [1.35 to 5.49]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 4.11 [1.25 to 5.49]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 4.78 [1.31 to 8.28]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 3.71 [1.31 to 4.27]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 1.41 [1.22 to 2.07]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 8.48 [1.31 to 15.41]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 3.52 [1.25 to 12.39]
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 1.68 [1.41 to 3.19]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 2.73 [1.38 to 4.07]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 1.22 [1.08 to 1.48]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 11.76 [3.22 to 37.22]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 4.07 [1.38 to 13.96]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 8.54 [4.07 to 13.67]
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 1.40 [1.08 to 9.72]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 2.76 [1.38 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 2.07 [1.22 to 4.14]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 3.12 [1.31 to 4.11]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 3.98 [1.18 to 16.92]

8. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP), based on RECIST v1.1, was defined as time from the first day of study treatment to the first occurrence of progressive disease or death due to disease progression, whichever occurred first. PD: At least a 20% increase in the sum of diameters of all target and all new measurable lesions.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 397
months
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 4.14 [1.31 to 8.34]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 3.45 [1.35 to 4.60]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 1.51 [0.72 to 10.97]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 2.73 [1.45 to 4.01]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 1.38 [0.99 to 1.54]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 1.51 [1.25 to 4.70]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 2.69 [1.28 to 3.12]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 1.41 [1.15 to 2.79]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 1.31 [1.25 to 1.35]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 2.73 [1.38 to 3.55]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 1.43 [1.25 to 14.39]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 2.96 [1.28 to 16.69]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 1.87 [1.35 to 5.49]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 4.11 [1.25 to 5.49]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 4.78 [1.31 to 8.28]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 3.71 [1.31 to 4.27]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 1.41 [1.22 to 2.07]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 8.48 [1.31 to 15.41]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 5.52 [1.25 to 23.33]
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 1.68 [1.41 to 3.19]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 2.73 [1.38 to 4.07]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 1.22 [1.08 to 1.48]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 12.58 [3.22 to 37.22]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 2.76 [1.38 to 13.86]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 8.54 [4.07 to 10.94]
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 1.40 [1.08 to 9.72]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 2.76 [1.38 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 2.07 [1.22 to 4.14]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 3.12 [1.31 to 4.11]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 3.98 [1.18 to 16.92]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first day of study treatment to death from any cause.
Time Frame: Baseline until death due to any cause (up to 4.5 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 397
months
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 14.78 [10.55 to 26.51]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 17.97 [8.90 to 27.56]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 6.41 [0.99 to 22.90]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 24.02 [4.11 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 5.09 [1.77 to 7.03]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 12.71 [4.37 to 24.44]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 9.66 [3.12 to 13.67]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 7.39 [2.89 to 11.70]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 5.59 [3.52 to 9.26]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 17.74 [6.37 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 8.33 [2.43 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 12.65 [2.50 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 21.98 [4.76 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 17.81 [9.10 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 12.78 [4.21 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 7.49 [3.25 to 11.20]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 4.62 [1.87 to 12.78]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | NA [NA to NA] — Median OS was not reached.
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 18.92 [3.52 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 8.57 [2.99 to 18.07]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 8.15 [6.14 to 16.49]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 8.39 [2.69 to 20.27]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | NA [NA to NA] — Median OS was not reached.
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | NA [NA to NA] — Median OS was not reached.
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 27.20 [17.02 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 16.16 [4.04 to 26.32]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 12.58 [2.40 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 15.52 [5.49 to NA] — Upper limit of CI was not reached due to low number of participants with events.
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | NA [NA to NA] — Median OS was not reached.
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 18.66 [1.41 to NA] — Upper limit of CI was not reached due to low number of participants with events.

10. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to 4.5 years
Population: Safety analysis set included all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 474
Participants | 435

11. Secondary Outcome: Treatment Duration of Atezolizumab
Time Frame: Baseline up to approximately 4.5 years
Population: Safety analysis set included all participants who received at least one dose of study medication.
Measure: Median (Full Range); unit: months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 474
months | 2.513 [0.03 to 52.47]

12. Secondary Outcome: Mean Number of Doses of Atezolizumab
Time Frame: Baseline up to approximately 4.5 years
Population: Safety analysis set included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Atezolizumab
Number analyzed (Participants) | 474
doses | 9.0 (11.28)

13. Secondary Outcome: Percentage of Participants With Anti-drug Antibodies (ADAs) to Atezolizumab
Time Frame: Baseline up to 4.5 years
Population: Safety analysis set included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 474
percentage of participants
  Baseline ADAs: number analyzed (Participants) | 462
  Baseline ADAs | 1.9
  Treatment-emergent ADAs: number analyzed (Participants) | 449
  Treatment-emergent ADAs | 18.3

14. Secondary Outcome: Serum Concentration of Atezolizumab
Time Frame: Predose and postdose on Day 1 of Cycle 1, predose on Day 1 of Cycles 2, 3, 4, 8 (cycle length = 21 days), and every 8 cycles until treatment discontinuation; at follow up (approximately 120 days after last dose) up to approximately 4.5 years
Population: Safety analysis set included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 474
ng/mL
  Cycle 01, Day 1 predose: number analyzed (Participants) | 452
  Cycle 01, Day 1 predose | 45528.4 (84303.42)
  Cycle 01, Day 1 postdose: number analyzed (Participants) | 454
  Cycle 01, Day 1 postdose | 422792.0 (225600.85)
  Cycle 02, Day 1 predose: number analyzed (Participants) | 433
  Cycle 02, Day 1 predose | 85674.3 (35394.34)
  Cycle 03, Day 1 predose: number analyzed (Participants) | 342
  Cycle 03, Day 1 predose | 131868.7 (60596.06)
  Cycle 04, Day 1 predose: number analyzed (Participants) | 288
  Cycle 04, Day 1 predose | 156555.7 (67478.76)
  Cycle 08, Day 1 predose: number analyzed (Participants) | 156
  Cycle 08, Day 1 predose | 201332.1 (96547.07)
  Cycle 16, Day 1 predose: number analyzed (Participants) | 72
  Cycle 16, Day 1 predose | 216038.7 (97136.92)
  Cycle 24, Day 1 predose: number analyzed (Participants) | 32
  Cycle 24, Day 1 predose | 224556.7 (104892.34)
  Cycle 32, Day 1 predose: number analyzed (Participants) | 21
  Cycle 32, Day 1 predose | 253873.7 (136820.70)
  Cycle 40, Day 1 predose: number analyzed (Participants) | 12
  Cycle 40, Day 1 predose | 284000.0 (110167.55)
  Cycle 48, Day 1 predose: number analyzed (Participants) | 8
  Cycle 48, Day 1 predose | 319500.0 (203543.61)
  Cycle 56, Day 1 predose: number analyzed (Participants) | 1
  Cycle 56, Day 1 predose | 203000.0 (NA) — Only 1 participant was analyzed at this time point.
  Cycle 64, Day 1 predose: number analyzed (Participants) | 2
  Cycle 64, Day 1 predose | 217000.0 (57982.76)
  Follow Up: number analyzed (Participants) | 77
  Follow Up | 17565.6 (29505.18)

15. Secondary Outcome: Percentage of Participants by Best Overall Response Based on Modified RECIST v1.1 (mBOR)
Description: Modified RECIST was based on the following: 1) New measurable lesions were added into the total tumor burden and followed; 2) Non-target lesions contributed only in the assessment of a CR; 3) Radiographic progression was determined only on the basis of measurable disease; had to be confirmed by a consecutive assessment =/>4 weeks from the date first documented. mBOR: 1) CR: overall tumor response assessment of CR at 2 consecutive visits at least 28 days apart. 2) PR: overall tumor response assessment of PR/CR at 2 consecutive visits at least 28 days apart without being a CR. 3) SD: overall tumor response assessment of SD/PR/CR at one or more visits at least 42 days after start of study treatment, but was not a confirmed CR or PR. 4) PD: an overall tumor response assessment of PD at any visit, and did not meet the criteria for a BOR of CR, PR or SD. 5) Missing: an assessment of SD, PR or CR in the first 42 days after start of study treatment and no further tumor assessments thereafter.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population: CR | 0.7
  Overall Population: PR | 7.2
  Overall Population: SD | 43.9
  Overall Population: PD | 38.3
  Overall Population: Missing | 9.9
  Cervical Cancer: CR: number analyzed (Participants) | 27
  Cervical Cancer: CR | 3.7
  Cervical Cancer: PR: number analyzed (Participants) | 27
  Cervical Cancer: PR | 11.1
  Cervical Cancer: SD: number analyzed (Participants) | 27
  Cervical Cancer: SD | 44.4
  Cervical Cancer: PD: number analyzed (Participants) | 27
  Cervical Cancer: PD | 25.9
  Cervical Cancer: Missing: number analyzed (Participants) | 27
  Cervical Cancer: Missing | 14.8
  Nasopharyngeal Carcinoma: CR: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: CR | 0
  Nasopharyngeal Carcinoma: PR: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: PR | 11.1
  Nasopharyngeal Carcinoma: SD: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: SD | 51.9
  Nasopharyngeal Carcinoma: PD: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: PD | 33.3
  Nasopharyngeal Carcinoma: Missing: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma: Missing | 3.7
  MSI-H or MMR Deficient Colorectal Cancer: CR: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: CR | 0
  MSI-H or MMR Deficient Colorectal Cancer: PR: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: PR | 0
  MSI-H or MMR Deficient Colorectal Cancer: SD: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: SD | 60.0
  MSI-H or MMR Deficient Colorectal Cancer: PD: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: PD | 30.0
  MSI-H or MMR Deficient Colorectal Cancer: Missing: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer: Missing | 10.0
  BRCA Mutated Ovarian Cancer: CR: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: CR | 0
  BRCA Mutated Ovarian Cancer: PR: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: PR | 13.3
  BRCA Mutated Ovarian Cancer: SD: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: SD | 40.0
  BRCA Mutated Ovarian Cancer: PD: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: PD | 33.3
  BRCA Mutated Ovarian Cancer: Missing: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer: Missing | 13.3
  BRCA Mutated Breast Cancer: CR: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: CR | 0
  BRCA Mutated Breast Cancer: PR: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: PR | 0
  BRCA Mutated Breast Cancer: SD: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: SD | 25.0
  BRCA Mutated Breast Cancer: PD: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: PD | 58.3
  BRCA Mutated Breast Cancer: Missing: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer: Missing | 16.7
  Liposarcoma: CR: number analyzed (Participants) | 13
  Liposarcoma: CR | 0
  Liposarcoma: PR: number analyzed (Participants) | 13
  Liposarcoma: PR | 0
  Liposarcoma: SD: number analyzed (Participants) | 13
  Liposarcoma: SD | 38.5
  Liposarcoma: PD: number analyzed (Participants) | 13
  Liposarcoma: PD | 53.8
  Liposarcoma: Missing: number analyzed (Participants) | 13
  Liposarcoma: Missing | 7.7
  Leiomyosarcoma: CR: number analyzed (Participants) | 17
  Leiomyosarcoma: CR | 0
  Leiomyosarcoma: PR: number analyzed (Participants) | 17
  Leiomyosarcoma: PR | 5.9
  Leiomyosarcoma: SD: number analyzed (Participants) | 17
  Leiomyosarcoma: SD | 23.5
  Leiomyosarcoma: PD: number analyzed (Participants) | 17
  Leiomyosarcoma: PD | 47.1
  Leiomyosarcoma: Missing: number analyzed (Participants) | 17
  Leiomyosarcoma: Missing | 23.5
  Gastrointestinal Stromal Tumor (GIST): CR: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): CR | 0
  Gastrointestinal Stromal Tumor (GIST): PR: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): PR | 0
  Gastrointestinal Stromal Tumor (GIST): SD: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): SD | 40.0
  Gastrointestinal Stromal Tumor (GIST): PD: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): PD | 60.0
  Gastrointestinal Stromal Tumor (GIST): Missing: number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST): Missing | 0
  Undifferentiated Pleomorphic Sarcoma: CR: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: CR | 0
  Undifferentiated Pleomorphic Sarcoma: PR: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: PR | 0
  Undifferentiated Pleomorphic Sarcoma: SD: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: SD | 9.1
  Undifferentiated Pleomorphic Sarcoma: PD: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: PD | 81.8
  Undifferentiated Pleomorphic Sarcoma: Missing: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma: Missing | 9.1
  Known Translocation-Related Sarcomas: CR: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: CR | 0
  Known Translocation-Related Sarcomas: PR: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: PR | 7.7
  Known Translocation-Related Sarcomas: SD: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: SD | 46.2
  Known Translocation-Related Sarcomas: PD: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: PD | 30.8
  Known Translocation-Related Sarcomas: Missing: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas: Missing | 15.4
  Radiation Induced Sarcoma: CR: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: CR | 0
  Radiation Induced Sarcoma: PR: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: PR | 12.5
  Radiation Induced Sarcoma: SD: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: SD | 37.5
  Radiation Induced Sarcoma: PD: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: PD | 37.5
  Radiation Induced Sarcoma: Missing: number analyzed (Participants) | 8
  Radiation Induced Sarcoma: Missing | 12.5
  Osteosarcoma: CR: number analyzed (Participants) | 11
  Osteosarcoma: CR | 0
  Osteosarcoma: PR: number analyzed (Participants) | 11
  Osteosarcoma: PR | 9.1
  Osteosarcoma: SD: number analyzed (Participants) | 11
  Osteosarcoma: SD | 36.4
  Osteosarcoma: PD: number analyzed (Participants) | 11
  Osteosarcoma: PD | 54.5
  Osteosarcoma: Missing: number analyzed (Participants) | 11
  Osteosarcoma: Missing | 0
  Chondrosarcoma: CR: number analyzed (Participants) | 12
  Chondrosarcoma: CR | 0
  Chondrosarcoma: PR: number analyzed (Participants) | 12
  Chondrosarcoma: PR | 0
  Chondrosarcoma: SD: number analyzed (Participants) | 12
  Chondrosarcoma: SD | 50.0
  Chondrosarcoma: PD: number analyzed (Participants) | 12
  Chondrosarcoma: PD | 41.7
  Chondrosarcoma: Missing: number analyzed (Participants) | 12
  Chondrosarcoma: Missing | 8.3
  Pleural Mesothelioma: CR: number analyzed (Participants) | 13
  Pleural Mesothelioma: CR | 0
  Pleural Mesothelioma: PR: number analyzed (Participants) | 13
  Pleural Mesothelioma: PR | 7.7
  Pleural Mesothelioma: SD: number analyzed (Participants) | 13
  Pleural Mesothelioma: SD | 61.5
  Pleural Mesothelioma: PD: number analyzed (Participants) | 13
  Pleural Mesothelioma: PD | 23.1
  Pleural Mesothelioma: Missing: number analyzed (Participants) | 13
  Pleural Mesothelioma: Missing | 7.7
  Peritoneal Mesothelioma: CR: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: CR | 0
  Peritoneal Mesothelioma: PR: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: PR | 14.3
  Peritoneal Mesothelioma: SD: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: SD | 50.0
  Peritoneal Mesothelioma: PD: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: PD | 14.3
  Peritoneal Mesothelioma: Missing: number analyzed (Participants) | 14
  Peritoneal Mesothelioma: Missing | 21.4
  Cholangiocarcinoma/Cancer of the Biliary Tract: CR: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: CR | 0
  Cholangiocarcinoma/Cancer of the Biliary Tract: PR: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: PR | 0
  Cholangiocarcinoma/Cancer of the Biliary Tract: SD: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: SD | 69.2
  Cholangiocarcinoma/Cancer of the Biliary Tract: PD: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: PD | 15.4
  Cholangiocarcinoma/Cancer of the Biliary Tract: Missing: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract: Missing | 15.4
  Anaplastic Thyroid Cancer (TC): CR: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): CR | 0
  Anaplastic Thyroid Cancer (TC): PR: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): PR | 0
  Anaplastic Thyroid Cancer (TC): SD: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): SD | 13.3
  Anaplastic Thyroid Cancer (TC): PD: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): PD | 73.3
  Anaplastic Thyroid Cancer (TC): Missing: number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC): Missing | 13.3
  Follicular or Papillary Thyroid Cancer (TC): CR: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): CR | 0
  Follicular or Papillary Thyroid Cancer (TC): PR: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): PR | 9.1
  Follicular or Papillary Thyroid Cancer (TC): SD: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): SD | 72.7
  Follicular or Papillary Thyroid Cancer (TC): PD: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): PD | 9.1
  Follicular or Papillary Thyroid Cancer (TC): Missing: number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC): Missing | 9.1
  Medullary/Follicular/Papillary TC: CR: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: CR | 0
  Medullary/Follicular/Papillary TC: PR: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: PR | 0
  Medullary/Follicular/Papillary TC: SD: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: SD | 42.9
  Medullary/Follicular/Papillary TC: PD: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: PD | 42.9
  Medullary/Follicular/Papillary TC: Missing: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC: Missing | 14.3
  Gastric/GE Junction Adenocarcinoma: CR: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: CR | 0
  Gastric/GE Junction Adenocarcinoma: PR: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: PR | 7.1
  Gastric/GE Junction Adenocarcinoma: SD: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: SD | 35.7
  Gastric/GE Junction Adenocarcinoma: PD: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: PD | 35.7
  Gastric/GE Junction Adenocarcinoma: Missing: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma: Missing | 21.4
  Malignant Germ Cell Tumors: CR: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: CR | 0
  Malignant Germ Cell Tumors: PR: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: PR | 0
  Malignant Germ Cell Tumors: SD: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: SD | 50.0
  Malignant Germ Cell Tumors: PD: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: PD | 50.0
  Malignant Germ Cell Tumors: Missing: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors: Missing | 0
  ER+/HER2- Hypermutated MBC: CR: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: CR | 0
  ER+/HER2- Hypermutated MBC: PR: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: PR | 8.3
  ER+/HER2- Hypermutated MBC: SD: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: SD | 25.0
  ER+/HER2- Hypermutated MBC: PD: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: PD | 58.3
  ER+/HER2- Hypermutated MBC: Missing: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC: Missing | 8.3
  Thymoma: CR: number analyzed (Participants) | 13
  Thymoma: CR | 0
  Thymoma: PR: number analyzed (Participants) | 13
  Thymoma: PR | 38.5
  Thymoma: SD: number analyzed (Participants) | 13
  Thymoma: SD | 46.2
  Thymoma: PD: number analyzed (Participants) | 13
  Thymoma: PD | 7.7
  Thymoma: Missing: number analyzed (Participants) | 13
  Thymoma: Missing | 7.7
  Thymic cancer: CR: number analyzed (Participants) | 12
  Thymic cancer: CR | 0
  Thymic cancer: PR: number analyzed (Participants) | 12
  Thymic cancer: PR | 8.3
  Thymic cancer: SD: number analyzed (Participants) | 12
  Thymic cancer: SD | 50.0
  Thymic cancer: PD: number analyzed (Participants) | 12
  Thymic cancer: PD | 33.3
  Thymic cancer: Missing: number analyzed (Participants) | 12
  Thymic cancer: Missing | 8.3
  Low/Intermediate Grade Carcinoid: CR: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: CR | 0
  Low/Intermediate Grade Carcinoid: PR: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: PR | 0
  Low/Intermediate Grade Carcinoid: SD: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: SD | 100.0
  Low/Intermediate Grade Carcinoid: PD: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: PD | 0
  Low/Intermediate Grade Carcinoid: Missing: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid: Missing | 0
  Poorly Differentiated Grade (excluding SCLC): CR: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): CR | 0
  Poorly Differentiated Grade (excluding SCLC): PR: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): PR | 16.7
  Poorly Differentiated Grade (excluding SCLC): SD: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): SD | 16.7
  Poorly Differentiated Grade (excluding SCLC): PD: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): PD | 58.3
  Poorly Differentiated Grade (excluding SCLC): Missing: number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC): Missing | 8.3
  Head and Neck Squamous Cell Carcinoma: CR: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: CR | 16.7
  Head and Neck Squamous Cell Carcinoma: PR: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: PR | 0
  Head and Neck Squamous Cell Carcinoma: SD: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: SD | 33.3
  Head and Neck Squamous Cell Carcinoma: PD: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: PD | 50.0
  Head and Neck Squamous Cell Carcinoma: Missing: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma: Missing | 0
  Penile Cancer: CR: number analyzed (Participants) | 4
  Penile Cancer: CR | 0
  Penile Cancer: PR: number analyzed (Participants) | 4
  Penile Cancer: PR | 0
  Penile Cancer: SD: number analyzed (Participants) | 4
  Penile Cancer: SD | 50.0
  Penile Cancer: PD: number analyzed (Participants) | 4
  Penile Cancer: PD | 50.0
  Penile Cancer: Missing: number analyzed (Participants) | 4
  Penile Cancer: Missing | 0
  Anal Cancer: CR: number analyzed (Participants) | 11
  Anal Cancer: CR | 9.1
  Anal Cancer: PR: number analyzed (Participants) | 11
  Anal Cancer: PR | 0
  Anal Cancer: SD: number analyzed (Participants) | 11
  Anal Cancer: SD | 45.5
  Anal Cancer: PD: number analyzed (Participants) | 11
  Anal Cancer: PD | 45.5
  Anal Cancer: Missing: number analyzed (Participants) | 11
  Anal Cancer: Missing | 0
  Known MSI High or MMR Deficient Tumors: CR: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: CR | 0
  Known MSI High or MMR Deficient Tumors: PR: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: PR | 20.0
  Known MSI High or MMR Deficient Tumors: SD: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: SD | 60.0
  Known MSI High or MMR Deficient Tumors: PD: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: PD | 20.0
  Known MSI High or MMR Deficient Tumors: Missing: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors: Missing | 0

16. Secondary Outcome: ORR Based on Modified RECIST v1.1
Description: Modified RECIST was based on the following: 1) New measurable lesions were added into the total tumor burden and followed; 2) Non-target lesions contributed only in the assessment of a CR; 3) Radiographic progression was determined only on the basis of measurable disease; had to be confirmed by a consecutive assessment =/>4 weeks from the date first documented. ORR was defined as the percentage of participants with CR or PR. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population | 7.9 [5.5 to 10.8]
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 14.8 [4.2 to 33.7]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 11.1 [2.4 to 29.2]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 0.0 [0.0 to 30.8]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 13.3 [1.7 to 40.5]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 0.0 [0.0 to 26.5]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 0.0 [0.0 to 24.7]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 5.9 [0.1 to 28.7]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 0.0 [0.0 to 21.8]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 0.0 [0.0 to 28.5]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 7.7 [0.9 to 25.1]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 12.5 [0.3 to 52.7]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 9.1 [0.2 to 41.3]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 0.0 [0.0 to 26.5]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 7.7 [0.2 to 36.0]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 14.3 [1.8 to 42.8]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 0.0 [0.0 to 24.7]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 0.0 [0.0 to 21.8]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 9.1 [0.2 to 41.3]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 0.0 [0.0 to 41.0]
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 7.1 [0.2 to 33.9]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 0.0 [0.0 to 23.2]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 8.3 [0.2 to 38.5]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 38.5 [13.9 to 68.4]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 8.3 [0.2 to 38.5]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 0.0 [0.0 to 26.5]
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 16.7 [2.1 to 48.4]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 16.7 [0.4 to 64.1]
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 0.0 [0.0 to 60.2]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 9.1 [0.2 to 41.3]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 20.0 [2.5 to 55.6]

17. Secondary Outcome: CBR Based on Modified RECIST v1.1
Description: Modified RECIST was based on the following: 1) New measurable lesions were added into the total tumor burden and followed; 2) Non-target lesions contributed only in the assessment of a CR; 3) Radiographic progression was determined only on the basis of measurable disease; had to be confirmed by a consecutive assessment =/>4 weeks from the date first documented. CBR was defined as the percentage of participants with CR, PR, or SD lasting for >/=6 weeks. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the diameters of all target and all new measurable lesions in the absence of CR. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD: At least a 20% increase in the sum of diameters of all target and all new measurable lesions.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 433
percentage of participants
  Overall Population | 51.7 [46.9 to 56.5]
  Cervical Cancer: number analyzed (Participants) | 27
  Cervical Cancer | 59.3 [38.8 to 77.6]
  Nasopharyngeal Carcinoma: number analyzed (Participants) | 27
  Nasopharyngeal Carcinoma | 63.0 [42.4 to 80.6]
  MSI-H or MMR Deficient Colorectal Cancer: number analyzed (Participants) | 10
  MSI-H or MMR Deficient Colorectal Cancer | 60.0 [26.2 to 87.8]
  BRCA Mutated Ovarian Cancer: number analyzed (Participants) | 15
  BRCA Mutated Ovarian Cancer | 53.3 [26.6 to 78.7]
  BRCA Mutated Breast Cancer: number analyzed (Participants) | 12
  BRCA Mutated Breast Cancer | 25.0 [5.5 to 57.2]
  Liposarcoma: number analyzed (Participants) | 13
  Liposarcoma | 38.5 [13.9 to 68.4]
  Leiomyosarcoma: number analyzed (Participants) | 17
  Leiomyosarcoma | 29.4 [10.3 to 56.0]
  Gastrointestinal Stromal Tumor (GIST): number analyzed (Participants) | 15
  Gastrointestinal Stromal Tumor (GIST) | 40.0 [16.3 to 67.7]
  Undifferentiated Pleomorphic Sarcoma: number analyzed (Participants) | 11
  Undifferentiated Pleomorphic Sarcoma | 9.1 [0.2 to 41.3]
  Known Translocation-Related Sarcomas: number analyzed (Participants) | 26
  Known Translocation-Related Sarcomas | 53.8 [33.4 to 73.4]
  Radiation Induced Sarcoma: number analyzed (Participants) | 8
  Radiation Induced Sarcoma | 50.0 [15.7 to 84.3]
  Osteosarcoma: number analyzed (Participants) | 11
  Osteosarcoma | 45.5 [16.7 to 76.6]
  Chondrosarcoma: number analyzed (Participants) | 12
  Chondrosarcoma | 50.0 [21.1 to 78.9]
  Pleural Mesothelioma: number analyzed (Participants) | 13
  Pleural Mesothelioma | 69.2 [38.6 to 90.9]
  Peritoneal Mesothelioma: number analyzed (Participants) | 14
  Peritoneal Mesothelioma | 64.3 [35.1 to 87.2]
  Cholangiocarcinoma/Cancer of the Biliary Tract: number analyzed (Participants) | 13
  Cholangiocarcinoma/Cancer of the Biliary Tract | 69.2 [38.6 to 90.9]
  Anaplastic Thyroid Cancer (TC): number analyzed (Participants) | 15
  Anaplastic Thyroid Cancer (TC) | 13.3 [1.7 to 40.5]
  Follicular or Papillary Thyroid Cancer (TC): number analyzed (Participants) | 11
  Follicular or Papillary Thyroid Cancer (TC) | 81.8 [48.2 to 97.7]
  Medullary/Follicular/Papillary TC: number analyzed (Participants) | 7
  Medullary/Follicular/Papillary TC | 42.9 [9.9 to 81.6]
  Gastric/GE Junction Adenocarcinoma: number analyzed (Participants) | 14
  Gastric/GE Junction Adenocarcinoma | 42.9 [17.7 to 71.1]
  Malignant Germ Cell Tumors: number analyzed (Participants) | 14
  Malignant Germ Cell Tumors | 50.0 [23.0 to 77.0]
  ER+/HER2- Hypermutated MBC: number analyzed (Participants) | 12
  ER+/HER2- Hypermutated MBC | 33.3 [9.9 to 65.1]
  Thymoma: number analyzed (Participants) | 13
  Thymoma | 84.6 [54.6 to 98.1]
  Thymic cancer: number analyzed (Participants) | 12
  Thymic cancer | 58.3 [27.7 to 84.8]
  Low/Intermediate Grade Carcinoid: number analyzed (Participants) | 12
  Low/Intermediate Grade Carcinoid | 100.0 [73.5 to 100.0]
  Poorly Differentiated Grade (excluding SCLC): number analyzed (Participants) | 12
  Poorly Differentiated Grade (excluding SCLC) | 33.3 [9.9 to 65.1]
  Head and Neck Squamous Cell Carcinoma: number analyzed (Participants) | 6
  Head and Neck Squamous Cell Carcinoma | 50.0 [11.8 to 88.2]
  Penile Cancer: number analyzed (Participants) | 4
  Penile Cancer | 50.0 [6.8 to 93.2]
  Anal Cancer: number analyzed (Participants) | 11
  Anal Cancer | 54.5 [23.4 to 83.3]
  Known MSI High or MMR Deficient Tumors: number analyzed (Participants) | 10
  Known MSI High or MMR Deficient Tumors | 80.0 [44.4 to 97.5]

ADVERSE EVENTS:
Time Frame: Up to approximately 4.5 years
Description: Safety analysis set included all participants who received at least one dose of study medication.
Arm/Group | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 310/474
Serious Adverse Events (participants affected / at risk) | 142/474
Other Adverse Events (participants affected / at risk) | 368/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=474)
ANAEMIA (Blood and lymphatic system disorders) | 8 (9)
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
LYMPH NODE HAEMORRHAGE (Blood and lymphatic system disorders) | 1 (1)
SPLENIC VEIN THROMBOSIS (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 (3)
GASTRIC ULCER (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2)
ILEUS (Gastrointestinal disorders) | 1 (1)
IMMUNE-MEDIATED ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 2 (2)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (2)
STOMATITIS (Gastrointestinal disorders) | 1 (1)
DEATH (General disorders) | 1 (1)
FATIGUE (General disorders) | 3 (3)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 (3)
MALAISE (General disorders) | 2 (2)
PYREXIA (General disorders) | 9 (9)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 1 (1)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1)
HEPATIC VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 2 (2)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1)
BILIARY TRACT INFECTION (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1)
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1)
ERYSIPELAS (Infections and infestations) | 2 (4)
HEPATITIS E (Infections and infestations) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 2 (2)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 (1)
MENINGITIS (Infections and infestations) | 1 (1)
PAROTITIS (Infections and infestations) | 1 (1)
PHARYNGITIS (Infections and infestations) | 2 (2)
PNEUMONIA (Infections and infestations) | 9 (9)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 4 (4)
SOFT TISSUE INFECTION (Infections and infestations) | 2 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 7 (9)
VIRAL INFECTION (Infections and infestations) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBELLAR ATAXIA (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 (3)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1)
DIPLEGIA (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 1 (1)
IMMUNE-MEDIATED ENCEPHALITIS (Nervous system disorders) | 1 (1)
MYASTHENIA GRAVIS (Nervous system disorders) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 2 (3)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1)
VAGINAL FISTULA (Reproductive system and breast disorders) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (8)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3)
TRACHEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
NEPHROSTOMY TUBE REMOVAL (Surgical and medical procedures) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1)
EMBOLISM (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=474)
ANAEMIA (Blood and lymphatic system disorders) | 59 (68)
HYPOTHYROIDISM (Endocrine disorders) | 37 (37)
ABDOMINAL PAIN (Gastrointestinal disorders) | 38 (44)
CONSTIPATION (Gastrointestinal disorders) | 46 (49)
DIARRHOEA (Gastrointestinal disorders) | 73 (86)
NAUSEA (Gastrointestinal disorders) | 68 (75)
VOMITING (Gastrointestinal disorders) | 56 (61)
ASTHENIA (General disorders) | 57 (61)
FATIGUE (General disorders) | 107 (112)
OEDEMA PERIPHERAL (General disorders) | 34 (34)
PYREXIA (General disorders) | 61 (73)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 25 (27)
WEIGHT DECREASED (Investigations) | 24 (24)
DECREASED APPETITE (Metabolism and nutrition disorders) | 67 (70)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 24 (25)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 31 (33)
MYALGIA (Musculoskeletal and connective tissue disorders) | 29 (33)
HEADACHE (Nervous system disorders) | 29 (34)
COUGH (Respiratory, thoracic and mediastinal disorders) | 44 (45)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 49 (50)
PRURITUS (Skin and subcutaneous tissue disorders) | 34 (46)
RASH (Skin and subcutaneous tissue disorders) | 40 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT02458638/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT02458638/SAP_001.pdf